CLINICAL TRIAL: NCT05923944
Title: Evaluating the Effect of Gamified Cognitive Training and of Casual Videogame Play on Anxiety in Adolescents: Protocol for a Randomized Controlled Trial
Brief Title: Video Game Play to Alleviate Adolescent Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other); University of Haifa (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10001C_212812
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Anxiety Disorders and Symptoms
Keywords: Digital mental health; Video Games; Cognitive Training; Emotion Regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eco-Rescue - Attentional Control - intervention (Experimental): The Eco-Rescue training intervention will be delivered through a dedicated video game installed on each participant's personal computer through the Steam platform, following a recommended training regimen of 30 minutes per day, 4 days per week for 6 weeks, for an expected total training duration of 12 hours.
  Interventions: Behavioral: Eco-Rescue
- Bejeweled 3 - Casual gaming - intervention (Experimental): The Bejeweled 3 training intervention will be delivered through a dedicated video game installed on each participant's personal computer through the Steam platform, following a recommended training regimen of 30 minutes per day, 4 days per week for 6 weeks, for an expected total training duration of 12 hours.
  Interventions: Behavioral: Bejelewed 3
- No-training intervention (No Intervention): The No-training intervention group does not involve any specific training program. Instead, participants assigned to this group will receive weekly phone calls, similar to the other groups, to answer the same questions as the other groups concerning their mental and emotional states and maintain regular contact throughout the 6-week study duration.

INTERVENTIONS:
Behavioral: Eco-Rescue — Ecorescue is a gamified adaptation of the multiple object tracking task (MOT) combined with a detection task. It requires to track the spatial position of specific moving targets among visually similar moving distractors, while at the same time detecting briefly flashed events. It was designed to load on attentional control and visuo-spatial working memory. Additionally, targets may express various facial emotions (happy, angry or neutral) requiring some emotional control in addition to attentional control.
  Arms: Eco-Rescue - Attentional Control - intervention
Behavioral: Bejelewed 3 — Bejeweled 3 is a commercially available puzzle video game developed and edited by PopCap Games. The main objective is to swap two adjacent gems of seven colors to create a line or row of 3 or more gems of the same type. When these gems are aligned, they disappear, and points are earned. The goal is to get as many points as possible until it is impossible to line up gems. Bejeweled 3 offers a variety of game modes that players can freely explore at their own pace, enhancing the overall enjoyment and providing increased variability during each gaming session. These game modes typically have shorter durations, with a single game usually lasting less than 5 minutes. Bejeweled 3 was chosen as it requires fewer attentional resources compared to Eco-Rescue and because it was reported to reduce stress and anxiety in adult samples (Russoniello et al. 2009, 2013).
  Arms: Bejeweled 3 - Casual gaming - intervention

SUMMARY:
Adolescence is a critical period for the onset and maintenance of anxiety disorders, which raises the importance of intervening early; one possibility of doing so is via digital interventions. At least two lines of research have been explored in the past years in this area. First, studies have tested the anxiolytic effects of casual video games, hypothesizing that, through the induction of flow, these games can effectively distract individuals from anxiety-related thoughts and feelings. Second, the bidirectional link between poor attentional control and higher anxiety has led to the design of novel interventions aiming to improve attentional control such as working memory training studies. Importantly, action video games, classified as a distinct gaming genre, have been shown to enhance attentional control. In this study, we aim to compare the effects of action video game play and casual game play to a no-training group, assessing their potential to alleviate anxiety when delivered entirely online. The goal of this three- arms randomized controlled trial is to evaluate the feasibility of a 6-week video game training intervention to reduce adolescent anxiety-related symptoms. We will also examine the efficacy of the proposed treatment when entirely deployed at adolescents' home.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 11-15 years
2. High-anxious score from the 41 items SCARED-Parent version (i.e. total score equal or above 17)
3. Access to a computer (at least Windows 7 or Mac OSX) at home and a reliable internet connection

Exclusion Criteria:

1. DSM diagnoses of Bipolar, Psychosis, Autism Spectrum Disorder, present or past.
2. Neurological injury (i.e. head injury)
3. Currently enrolled in another cognitive training intervention

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety assessed through the Screen for Child Anxiety Related Emotional Disorders Child Version (SCARED-C; Birmaher et al. 1999) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The SCARED-C is a 41 items self-report anxiety questionnaire with subscales measuring General Anxiety Disorder, Social Phobia Disorder, Panic Disorder, Separation Anxiety Disorder and School Avoidance. Participants are asked to rate each statement, referring to the past four weeks, on a scale ranging from 0 (Not True or Hardly Ever True) to 2 (Very True or Often True). A score of 25 or higher may indicate the presence of an Anxiety Disorder. Analysis of primary outcome will be based on this total score.

SECONDARY OUTCOMES:
Attentional Control assessed through the Useful Field of View Task (UFOV; Yung et al., 2015) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The UFOV is a computerized divided attention task where participants have to identify whether a briefly flashed smiley presented at the center of the screen has short or long hair and detect on which of the eight cardinal directions was a peripheral target stimulus presented, while ignoring other distractors. The presentation time is made shorter (more difficult) or longer (less difficult) according to a 3-down-1-up staircase. The task stops after 8 reversals or 72 trials, whichever happens first. Performance is measured by the mean presentation time of the last 5 trials (expressed in milliseconds). The task measures the efficiency of divided visual attention in the presence of visual distractors.
Attentional Control assessed through an adaptation of the Test of Variables of Attention (TOVA) as implemented in the ACE-X battery (Mars-UFO and Venus-UFO; https://neuroscape.ucsf.edu/researchers-ace/) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The TOVA is a computerized task where participants press a response key when presented with a visual stimulus in the upper part of the screen (go trials) and refrain from responding if flashed in the lower part of the screen (no-go trials). A first block evaluates sustained attention and a second impulsivity. In the sustained attention, go trials represent 25% of the trials; in the impulsivity block, go trials represent 75% of the trials.
Attentional Control assessed through the Multiple Objects Tracking Task (MOT; Yung et al., 2015) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The MOT is a computerized task in which participants are presented 16 yellow smileys moving freely within a circular area. During the first two seconds of each trial, a subset of these items is flagged as targets by being blue. Participants are instructed to track these blue smileys even though they turn back to yellow and become indistinguishable from the other items. After a few seconds, the items stop moving, one item is highlighted, and participants respond whether this item was initially flagged blue or not. MOT performance is measured as the percentage of correct responses (i.e. accuracy) in trials with 3, 4, 5 and 6 targets independently and combined overall. Higher accuracy score indicates better task performance. This task requires not only selecting targets amongst distractors but also dividing one's attention among these moving targets. Furthermore, it requires sustaining attention for a few seconds, necessitating both sustained attention and visuo-spatial working memory.
Affective Control assessed through the Affective Backward Digit Span Task (ABDS; modified version of Schweizer et al. 2019) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The ABDS is a computer-based task where participants are presented with digits (for 1500 ms) one after the other, and asked to recall them in reverse order. These are presented on a background of either neutral or affective images, in two different blocks, to manipulate valence. The images are sourced from the Geneva Affective Picture Database. In each trial, participants are presented with a series of single digits [0-9]. The length of the series to recall is increased or decreased by one digit depending on previous trial performance according to a 1-up-1-down staircase. No feedback is provided. After two reversals the block stops. Span is estimated for each block as the maximum correct length recalled. The span difference between the neutral versus affective blocks is an index of the individual ability to implement control in the face of affective distraction

OTHER OUTCOMES:
Emotion Regulation habits assessed through the Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski et al., 2001) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)]
  The CERQ is a 36-item self-report measure that captures stable-dispositional cognitive emotion regulation strategies when people experience stressful or threatening life experiences. Specifically, the following strategies are measured: Self-blame, blaming others, acceptance, refocusing on planning, positive refocusing, rumination, positive reappraisal, putting into perspective, and catastrophizing. Each subscale comprises 4 items and uses a 5-point scale (1 = almost never, 5 = almost always); the range of scores for each subscale is 4-20. Analysis of change will be based on the total score. A higher score represents greater use of cognitive coping strategies.
Subjective Attentional Control assessed through the Attention Control Scale (ACS; Derryberry et al., 2002). | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The ACS is a 20-item self-report questionnaire designed to measure the construct of attention focusing and attention shifting. 20 items are rated on a 4-point Likert Scale from 1 (almost never) to 4 (always). Respondents rate items according to their experience in the past 4 weeks. Analysis of change will be based on the total score and on scores of each subscale. A lower score indicates higher attentional control abilities.
Depressive symptoms assessed though the modified 8-item version of the Patient Health Questionnaire (PHQ-8; Kroenke et al., 2009) | Change from baseline (T1) at 1 week after training completion (T2), and at 4 months after training completion (T3)
  The PHQ-8 is designed to assess symptoms of depression. Participants are asked to indicate the frequency of experiencing eight specific problems or symptoms over the course of the past four weeks. (e.g., "feeling down, depressed, or hopeless," "feeling tired or having little energy,"). Each item is rated 0 (not at all), 1 (several days), 2 (more than half the days), or 3 (nearly every day). Analysis of change will be based on the total score. A higher score indicates higher depressive symptoms.
Sleep and Mood assessed through stand-alone questions for the duration of the training once a week. | Over the intervention period (4 weeks up to 8 weeks)
  Sleep: "During the past week, how would you rate your sleep quality overall. This question is rated from 1 (very poor) to 5 (very good).
  Positive mood: "How much have you experienced positive mood in the past week?" This question is rated from 1 (not at all) to 5 (extremely).
  Negative mood: "How much have you experienced negative mood in the past week?" This question is rated from 1 (not at all) to 5 (extremely).
Worry assessed with the following statement for the duration of the training once a week. | Over the intervention period (4 weeks up to 8 weeks)
  "During the past week I worried a lot." This item is rated 0 (not true), 1 (somewhat true), or 2 (true), and was taken from the Strengths and Difficulties Questionnaire (item 8 from the emotional problems scale, Goodman et al. 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Daphné Bavelier, Professor, Principal Investigator — University of Geneva, Switzerland; Swann Pichon, Professor, Principal Investigator — HES - Geneva School of Health Science, Switzerland; Tomer Shechner, Professor, Principal Investigator — University of Haifa, Israel
Locations (2):
- University of Haifa, Haifa, Israel
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hisamura M, Murao M. [Studies on the changes of vital functions during upper gastrointestinal endoscopy in the aged patients (author's transl)]. Nihon Ronen Igakkai Zasshi. 1981 Nov;18(6):469-75. No abstract available. Japanese. PMID 7339086
- [Background] Yung A, Cardoso-Leite P, Dale G, Bavelier D, Green CS. Methods to test visual attention online. J Vis Exp. 2015 Feb 19;(96):52470. doi: 10.3791/52470. PMID 25741746
- [Background] Schweizer S, Leung JT, Kievit R, Speekenbrink M, Trender W, Hampshire A, Blakemore SJ. Protocol for an app-based affective control training for adolescents: proof-of-principle double-blind randomized controlled trial. Wellcome Open Res. 2019 Oct 2;4:91. doi: 10.12688/wellcomeopenres.15229.2. eCollection 2019. PMID 31289755
- [Background] Pylyshyn ZW, Storm RW. Tracking multiple independent targets: evidence for a parallel tracking mechanism. Spat Vis. 1988;3(3):179-97. doi: 10.1163/156856888x00122. PMID 3153671
- [Background] Russoniello CV, O'Brien K, Parks JM. EEG, HRV and Psychological Correlates while Playing Bejeweled II: A Randomized Controlled Study. Stud Health Technol Inform. 2009;144:189-92. PMID 19592761
- [Background] Russoniello CV, Fish M, O'Brien K. The Efficacy of Casual Videogame Play in Reducing Clinical Depression: A Randomized Controlled Study. Games Health J. 2013 Dec;2(6):341-6. doi: 10.1089/g4h.2013.0010. Epub 2013 Nov 8. PMID 26197075
- [Background] Derryberry D, Reed MA. Anxiety-related attentional biases and their regulation by attentional control. J Abnorm Psychol. 2002 May;111(2):225-36. doi: 10.1037//0021-843x.111.2.225. PMID 12003445
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Garnefski, N., Kraaij, V., & Spinhoven, P. (2001). Negative life events, cognitive emotion regulation and emotional problems. Personality and Individual differences, 30(8), 1311-1327.
- [Background] Goodman R, Meltzer H, Bailey V. The Strengths and Difficulties Questionnaire: a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry. 1998 Sep;7(3):125-30. doi: 10.1007/s007870050057. PMID 9826298
- [Derived] Gradi N, Chopin A, Bavelier D, Shechner T, Pichon S. Evaluating the effect of action-like video game play and of casual video game play on anxiety in adolescents with elevated anxiety: protocol for a multi-center, parallel group, assessor-blind, randomized controlled trial. BMC Psychiatry. 2024 Jan 19;24(1):56. doi: 10.1186/s12888-024-05515-7. PMID 38243201
- See also: adaptation of the TOVA as implemented in the ACE-X battery — https://neuroscape.ucsf.edu/researchers-ace/